CLINICAL TRIAL: NCT04936074
Title: Comparison of Posterior Muscle-preserving Selective Laminectomy and Laminectomy With Fusion for Treating Degenerative Cervical Myelopathy: Myelopathy Randomized Controlled Trial (MyRanC)
Brief Title: Fusion or no Fusion After Decompression of the Spinal Cord in Patients With Degenerative Cervical Myelopathy
Acronym: MyRanC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Collaborators: Karolinska Institutet (Other); Linkoeping University (Other Government); Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Anna Mac Dowall, Consultant, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uppsala2021
Record Dates: First submitted 2021-05-19; First posted 2021-06-23 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Cervical Spondylotic Myelopathy
Keywords: Cervical fusion; Cervical spine; Laminectomy; Spinal surgery; Randomized controlled trial
MeSH Terms: conditions — Klippel-Feil Syndrome | interventions — Laminectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Muscle preserving selective laminectomy (L-group) (Experimental): Muscle-preserving selective laminectomy with a posterior midline incision and dissection through the nuchal fascia. The spinous processes are split in the midline using a high-speed burr/ultrasound knife and without disturbing the deep extensor muscles on either side. Angulating away from the midline, the spinous processes are divided at their bases. Laminectomy is performed with a width no more than 2-3 mm wider than the dural borders. The facet joints are not exposed. Finally, the split spionous processes are sutured together. No collar or restrictions will be used in either group.
  Interventions: Procedure: Muscle preserving selective laminectomy
- Laminectomy with instrumented fusion (LF-group) (Active Comparator): Laminectomy with instrumented fusion with a midline incision over the appropriate levels defined as the same levels as the extension of laminectomy plus one level above and below but not extending beyond C3-C7. Soft tissue dissection and retraction is performed to identify osseous landmarks. Special care is taken to spare muscle attachments on C2 and C7. Spinal instrumentation is performed with lateral mass or pedicle screws (C3-C7) combined with rod fixation. Laminectomy is performed with a width not extending more than 2 mm outside the dural borders. Facet joint injury should be avoided. Special care is taken to spare the C7 spinous process and distal half of C7 lamina. The sagittal alignment is corrected before spinal fixation. No collar or restrictions will be used in either group.
  Interventions: Procedure: Laminectomy with instrumented fusion

INTERVENTIONS:
Procedure: Muscle preserving selective laminectomy — Muscle-preserving selective laminectomy differ from traditional laminectomy by the spinous process split that preserves the deep extensor muscles. The bilateral facet joints are not exposed. After the laminectomy is finished the split fragments of the spinous process are sutured together so that the deep extensor muscles are restored.
  Arms: Muscle preserving selective laminectomy (L-group)
Procedure: Laminectomy with instrumented fusion — A traditional laminectomy is complemented with lateral mass and/or pedicle screws connected with rods.
  Arms: Laminectomy with instrumented fusion (LF-group)

SUMMARY:
Background:

Degenerative cervical myelopathy (DCM) is characterized by neck pain, neck stiffness, weakness, paresthesia, sphincter disturbance and balance disorder. The mean age for symptoms is 64 years and more men than women, 2.7:1, are affected. The most common level is C5-C6. DCM is the predominant cause of spinal cord dysfunction in the elderly worldwide. Surgical options include stand-alone laminectomy, laminectomy and fusion and laminoplasty. The preferable surgical approach is though, a matter of controversy. The objective of this study is to compare stand-alone laminectomy to laminectomy and fusion.

Methods/Design:

This is a multicenter randomized, controlled, parallel group non-inferiority trial. A total of 300 adult participants are allocated in a ratio of 1:1. The primary endpoint is reoperation for any reason within 5 years of follow-up. Sample size and power calculations were performed by estimating the reoperation rate after laminectomy to 3.4% and after laminectomy with fusion to 7.9% based on data from the Swedish spine registry (Swespine) on patients with DCM.

Secondary outcomes are the patient derived modified Japanese orthopaedic association (P-mJOA) score, Neck disability index (NDI), European quality of life five dimensions (EQ-5D), Numeric rating scale (NRS) for neck and arm pain, Hospital anxiety and depression scale (HADS), development of kyphosis measured as the cervical sagittal vertical axis (cSVA) and, death. Clinical and radiological follow-up is performed at 3, 12, 24 and 60 months after surgery. The main inclusion criteria is 1-4 levels of DCM in the subaxial spine, C3-C7, with or without deformity. The REDcap will be used for safe data management. Data will be analyzed in the per protocol (PP) population, defined as randomized patients who are still alive without having emigrated or left the study after five years.

Discussion:

This will be the first randomized controlled trial comparing two of the most common surgical treatments for DCM; the posterior muscle-preserving selective laminectomy and posterior laminectomy with instrumented fusion. The results of the MyRanC study will provide surgical treatment recommendations for DCM. This may result in improvements in surgical treatment and clinical practice regarding DCM.

DETAILED DESCRIPTION:
Background:

Degenerative cervical myelopathy (DCM) is characterized by neck pain and stiffness, weakness and paresthesia of the extremities, sphincter disturbance and bowel and balance disorder. DCM is the most common cause of spinal cord dysfunction in the elderly worldwide (1) and the incidence is 41 per million within North America (2). The mean age for symptoms is 64 years of age, more men than women, 2.7:1, are affected and the most common level is C5-C6 (3).

Mechanism:

DCM is typically the consequence of degenerative disc herniation, osteophyte formation and hypertrophy of the ligamentum flavum that compress the spinal cord. Ossification of the posterior longitudinal ligament (OPLL), which is more prevalent in the Asian population, may also cause compression of the spinal cord.

With non-operative treatments, i.e. medication and physiotherapy, 20-60% of the patients deteriorate neurologically and surgical treatment is indicated (4).

Existing knowledge:

The surgical treatment for DCM is decompression of the spinal cord. Decompression may be achieved with an anterior or posterior approach. Several algorithms have been proposed on whether to choose anterior diskectomy and fusion, anterior corpectomy and fusion, posterior laminectomy with fusion, posterior laminoplasty or, posterior laminectomy alone (5,6). Anterior discectomy/corpectomy with fusion is recommended in patients with a straight or kyphotic spine with compression of less than three levels (6). A posterior approach is recommended in patients with cervical lordosis and compression of more than three levels (7). The WFNS Spine Committee modified these recommendations in 2019 towards a wider use of posterior approaches, e.g. in patients with posterior compression at 1 or 2 levels and patients with a flexible kyphosis (8). It was recommended to address anterior compression with an anterior approach and posterior compression by a posterior approach. Hence, when propensity score matching is performed on the basis of MRI classification and description of the degenerative changes in each patient, anterior and/or posterior compression of the spinal cord, there is no difference between anterior or posterior decompression and fusion approaches (9).

Fusion is recommended in patients with DCM and concurrent signs of instability but there is no definition of instability in the degenerated cervical spine (10). In the traumatic cervical spine, however, instability is defined as >3.5 mm translation or 11° rotation on lateral flexion-extension radiographs (11) but there are no indications that degenerative changes with intact ligaments and unfractured joints would be unstable in the same way.

Kyphosis of cSVA > 40 mm (13) has been correlated to worse postoperative outcome (normal cSVA = 17-11 mm) (14). Consequently the recommendation is to correct kyphosis by an anterior approach (8) but a correction does not seem to affect the outcomes (15).

It remains a matter of debate among spinal surgeons whether posterior fusion after laminectomy for DCM, should be mandatory or not. After reports of post-laminectomy kyphosis in the 1970s and 1980s (16) prophylactic fusion has commonly been combined with the laminectomy procedure (9). In a report from 1999, 34% of the patients developed kyphosis or swan neck deformity after laminectomy compared with 7% of patients surgically treated with laminoplasty, using a muscle-preserving technique (17). However, a muscle-preserving technique that retains the facet integrity as well as the extensor musculature may be used when performing posterior laminectomy as well and is observed to maintain sagittal balance after surgery without progression of kyphosis (18).

Distal junction kyphosis (DJK) is a kyphotic angulation of at least 10° at the distal segment adjacent to a fused level and occurs in 24% of patients within a year after fusion surgery (19). Adjacent segment pathology (ASP) is progression of degeneration at the levels adjacent to a fused level and may also necessitate reoperation with decompression and extended fusion surgery (20).

Considering the existence of muscle-preserving laminectomy techniques that can maintain cervical lordosis (26), there is reason to explore the additional value of instrumented fusion in the cervical spine.

Although both methods are widely used, they are yet to be compared in a randomized controlled study.

Need for a trial:

There exists a controversy among spinal surgeons regarding the need for posterior fusion when laminectomy for DCM is performed.

We hypothesize that laminectomy without fusion results in shorter hospital stay and quicker return to an active life, without reduced patient satisfaction, functional scores, or delayed kyphosis.

It is important to achieve good outcome with a single surgery, to spare this frail group of patients from reoperations. Therefore, reoperation for any reason within five years after the primary surgery will be the primary endpoint of the current study. Long-term follow-up radiographs and magnetic resonance imaging (MRI) is needed to assess differences in the subsequent degenerative changes including spondylolisthesis, kyphosis, and adjacent segment pathology (ASP) to compare the two strategies.

Additionally, data from this study can be used to identify risk factors for poor outcome to guide surgical decision making.

Objectives:

* To determine the surgical treatment associated with the lowest frequency of reoperations when treating participants with CSM by performing a non-inferiority study comparing laminectomy alone with laminectomy and fusion.
* To evaluate potential differences in outcome including participant satisfaction, functional scores, late degenerative changes including spondylolisthesis, kyphosis, DJK, ASP and, death.

Study setting:

* Uppsala University Hospital
* Karolinska University Hospital, Stockholm
* Ryhov Hospital, Jönköping
* Sahlgrenska University Hospital, Gothenburg

Sample size:

Based on data from the national Swedish spine registry on patients with CSM, reoperation was estimated to 3.4% after standalone laminectomy and 7.9% after laminectomy and fusion. Five year mortality was estimated to 16.3% in the same population.

We further determined that excluding a 5% excess rate of reoperation in the laminectomy group vs laminectomy and fusion was a clinically relevant target for the study, and therefore set the non-inferiority margin at 5 percentage points (pp).

With a sample size of 300 participants and with regards to mortality and an additional 5% loss due to dropout and emigration, we end up with 236 analyzable patients. This results in a power of 87% based on simulation using rerandomization.

Recruitment:

All participants diagnosed with DCM referred for surgical consultation to the orthopedic or neurosurgery departments at the participating centers will be eligible for the study. Oral and written information about the study will be given at the routine physiotherapist appointment before the scheduled doctor's appointment and repeated by the treating surgeon at the following consultation. Participants may be enrolled if they meet the inclusion criteria and sign informed consent.

Allocation:

Participants will be allocated to either standalone laminectomy or laminectomy and fusion through randomization with a 1:1 ratio using the REDcap software (Research Electronic Data Capture), after informed consent and agreement to be included in the study. After inserting the patient´s personal number into REDcap the program reports the random allocation of the patient according to the pre-constructed randomization list. The randomization is stratified for center and participant sex, i.e. using separate lists for each center and sex. The allocation sequence utilizes balanced blocks of three different sizes occurring in random sequence. The principal investigator and study collaborators are blinded to the sequence, the block sizes and block sequence.

Blinding:

Trial participants will not be blinded after assignment to interventions as they have online access to their medical records by a centrally managed system.

The outcome assessors and data analysts will be blinded by using a coding system for the treatment groups.

Dropouts:

Dropouts may be one out of two entities; 1) the participant actively leaves the study or, 2) the participant has died or do not show up on follow-ups for unclear reasons. In case 1, the participant will not be part of the study anymore and data will not be retrieved from other information sources. In case 2, information about living participants will be retrieved from the medical records, radiographs, and the Swedish patient registry.

Statistical methods:

To test for non-inferiority, a two-sided 95% confidence interval (CI) for the difference in failure rates between the two groups will be computed. To account for sparsity of events, the CI will be computed using rerandomization techniques,10 blocked on sex, since the randomization was stratified on sex. Non-inferiority will be claimed if the upper limit of the CI is less than 5 pp. If non-inferiority is demonstrated, superiority will also be tested using the same CI, although the study is likely underpowered to detect this.

All endpoints will be analyzed in the per protocol (PP) population, defined as randomized patients who are still alive without having emigrated or left the study after five years.

The secondary outcomes listed above will be analyzed using ordinal regression models, adjusted for sex. In addition, each secondary endpoint will be dichotomized and analyzed using logistic regression. The dichotomization will be done by comparing baseline and follow-up data, either based on MCID when applicable, or else by defining success as an improvement from baseline. All secondary endpoints will be analyzed at 1, 2 and 5 years of follow-up, but not until the study is closed and the primary results is published.

The study statistician is Lars Lindhagen at Uppsala Clinical Research Center.

Data collection:

Questionnaires including baseline questionnaires and postal follow-up questionnaires as well as validated PROMs will be distributed the participants preoperatively. Postoperatively the participants are routinely followed via the Swespine (swespine.se) and follow-up questionnaires and PROMS will be retrieved from Swespine.41,49,50

Closing statement:

Degenerative cervical myelopathy is the most common cause of spinal cord dysfunction in the elderly worldwide and the incidence is 41 per million within North America. Until now there is no consensus whether to fuse or not when laminectomy is performed and the choice of surgical method is mainly up to the surgeon's preference.

This will be the first randomized controlled trial comparing two of the most common surgical treatments for DCM; the posterior muscle-preserving selective laminectomy and posterior laminectomy with instrumented fusion.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* 1-4 levels of cervical degenerative myelopathy in the subaxial spine, C3-C7, without or with deformity not exceeding exclusion criteria, see below.
* Eligible for both treatments
* Ability to understand and read Swedish language
* Symptomatic myelopathy with at least one clinical sign of myelopathy
* No previous spine surgery
* Psychosocially, mentally, and physically able to fully comply with this protocol, including adhering to scheduled visits, treatment plan, completing forms, and other study procedures
* Personally, signed and dated informed consent document prior to any study-related procedures, indicating that the patient has been informed of all pertinent aspects of the trial

  * Definition of kyphosis - cSVA > 40 mm and/or C2-C7 Cobb > 10° kyphosis. Definition of spondylolisthesis - anterior slippage of > 2 mm on cervical radiographs taken in the neutral position.

Exclusion Criteria:

* Local kyphosis; a modified K-line minimum interval distance (INT) of <4 mm
* Spondylolisthesis >4 mm and simultaneous translation >2 mm on lateral flexion/extension radiographs
* Soft disc herniations only (no signs of osteophyte formation and hypertrophy of the ligamentum flavum)
* Active infection
* Neoplasm
* Trauma
* Inflammatory disease (i.e., rheumatoid arthritis or ankylosing spondylitis or DISH)
* Systemic disease including HIV
* Lumbar or thoracic spinal disease to the extent that surgical consideration is probable or anticipated within 6 months after the cervical surgical treatment (significant lumbar stenosis as defined by Schizas C or worse).
* OPLL
* Parkinson´s disease
* Drug abuse, dementia, or other reason to suspect poor adherence to follow-up
* Previous cervical spine surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2030-02-01 (Estimated); Study Completion 2033-02-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be reoperation for any reason to reflect whether laminectomy alone or laminectomy with instrumented fusion results in fewer reoperations without increasing the frequency of complications. | Recorded at 5 years of follow-up
  Reoperation will be considered in case of:
  * Postoperative hematoma or reperfusion injury with neurologic deterioration within hours/days after the primary surgery.
  * Change in sagittal alignment (kyphosis, DJK of more than 40 mm cSVA and/or C2-C7 Cobb < -10°) with corresponding symptoms of camptocormia/increased pain/neurological deterioration.
  * ASP defined as degenerative changes on an adjacent level diagnosed with MRI and concomitant symptoms of myelopathy and/or radiculopathy.
  * Implant failure (clear radiolucency around >1 screw or rod breakage with increased neck pain and/or neurologic deterioration).
  * Postoperative infection that requires revision surgery.

SECONDARY OUTCOMES:
Change from baseline in myelopathy score on the patient derived modified Japanese Orthopedic Association scale (P-mJOA) at 2 years. | Measured at baseline and 2 years of follow-up
  P-mJOA is a self-administered questionnaire with four domains, measuring motor (upper and lower extremities), sensor (upper extremities) and sphincter dysfunction in patients with cervical degenerative myelopathy. The first domain is scored from zero to five, second domain from zero to seven, third and four domains from zero to three. The maximum score is 18 points, indicating no deficits and the minimum score is zero, total tetraplegia. The minimum clinically important difference (MCID) in mJOA has been reported to be 2 overall with a threshold of 1 in mild myelopathy (mJOA >14), 2 in moderate myelopathy (mJOA 12-14) and 3 in severe myelopathy (mJOA <12). Consistency between P-mJOA and mJOA is demonstrated with identical mean scores and a SD of 1.5 together with a strong agreement of 0.83 with the use of intraclass correlation coefficient and the Spearman correlation.
Change from baseline in participants disability score on the Neck disability index (NDI) at 2 years. | Measured at baseline and 2 years of follow-up
  Change of at least 17% in the NDI (100 points) compared with baseline (adjustable according to results from own minimal clinically important change results for Neck Disability Index).
  The NDI range from 0-100% with higher scores indicating severe disability. The MCID is 15%-17% for NDI.
Change from baseline in myelopathy score on the Nurick scale at 2 years. | Measured at baseline and 2 years of follow-up
  A six grade system (0-5) based on the 'difficulty in walking'.
Change from baseline in the patient Quality of life five dimensions (EQ-5D index) at 2 years. | Measured at baseline and 2 years of follow-up
  EQ-5D index range from -0.5 to 1 with higher scores reflecting a better quality of life).
Change from baseline in pain scores on the Numeric rating scale (NRS) at 2 years. | Measured at 2 years of follow-up
  Change in pain, as defined by ≥2.5 points on a 10 graded Numeric rating scale (NRS) for arm/shoulder pain.
  NRS for neck and arm pain range from 0-10, with higher scores indicating more severe pain. The MCID is 2.59 for NRS of the neck and arm.
Change at baseline in number of participants with psychological impairment on the Hospital anxiety and depression scale (HADS) in both groups. | Measured at baseline
  HADS range from 0-42 with higher scores indicating more anxiety/depression. The cutoff for depression defined as >10 p.
Change in number of satisfied participants on the patient global assessment in both groups at 2 years. | Measured at baseline and 2 years of follow-up
  The Global Assessment is a "satisfaction index" for evaluating the participants´ experienced overall result after surgery. The participant is asked "How is your attitude regarding the treatment result". The alternative answers are "satisfied", "uncertain", "dissatisfied".
Change from baseline in myelopathy on the 10-s grip and release test at 2 years. | Measured at baseline and 2 years of follow-up
  The 10-s grip and release test is performed with the forearm in pronation and the wrist in mild extension. The participant is asked to grip and release with their fingers as rapidly as possible and the number of completed cycles of movement within 10 seconds is counted.
Change from baseline in myelopathy on the 10-s foot-tapping speed test at 2 years. | Measured at baseline and 2 years of follow-up
  The 10-s foot-tapping speed test is performed with the participant sitting on a chair adjusted so that the hip and knee are flexed at 90° and the bilateral soles have contact with the floor. The participant is asked to move their toes up and down, tapping the floor as quickly as possible for 10 sec with their heels firmly planted on the floor. The number of completed cycles of movement within 10 seconds is counted.
Difference in number of participants with treatment-related adverse events in both groups at 5 years. | Recorded at 5 years of follow-up
  All adverse events in both groups will be presented. The adverse events will be graded according to severity: grade 1, any non-life-threatening complication treated without invasive procedures; grade 2, complications requiring invasive management such as surgical, endoscopic, and endovascular procedures; grade 3, life-threatening adverse events requiring treatment in an intensive care unit (ICU); and grade 4, deaths as a result of complications.
Change from baseline in sagittal alignment on neutral radiographs at 5 years. | Assessed preoperatively and at 5 years of follow-up
  Standing radiographs of the cervical spine in neutral, flexion and extension will be performed. When radiographs of the neutral position are executed the patient will be in a comfortable standing position with the head facing forward for horizontal gaze. The radiographs will be used to investigate the sagittal alignment by measuring the C2-C7 Cobb angle, C2-C7 sagittal vertical axis (cSVA), C7 slope and T1 slope.
Number of participants with change in adjacent segment pathology (ASP) on MRIs from baseline to 5 years of follow-up. | Assessed preoperatively and at 5 years of follow-up
  Magnetic resonance imaging (MRI) of the cervical spine with T1- and T2-weighted images in sagittal and T2-weighted in axial planes will be performed. Hereby the degenerative development over time may be assessed.
Number of participants with change in compression of the spinal cord on the index level on MRIs from baseline to 5 years of follow-up. | Assessed preoperatively and at 5 years of follow-up
  Magnetic resonance imaging (MRI) of the cervical spine with T1- and T2-weighted images in sagittal and T2-weighted in axial planes will be performed preoperatively, after three months and at five years of follow-up. Hereby the compression of the spinal cord may be assessed as well as the performed decompression and the degenerative development over time.
Change in direct costs between the groups at 1 year of follow-up. | Recorded at 1 year of follow-up.
  Direct costs includes hospital stay related to the surgical procedure, implant related costs, and pain medication usage.
Change in indirect societal costs at one years of follow-up. | Recorded at 1 year of follow-up
  Indirect costs includes pain medication usage, societal costs for absence from work and workers compensation.
Mortality | Recorded at 5 years of follow-up
  Death and cause of death will be recorded within the study.

CONTACTS AND LOCATIONS:
Overall Officials: Anna MacDowall, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Academic Hospital of Uppsala, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
The REDcap* with a two-stage verification login will be used for safe data management. Participants will be coded, and collaborators and statisticians will only have access to encrypted data. Access to decrypted data and safekeeping of the decryption key will be limited to the principal investigator and the study nurse. Participating spine surgeons have only access to his/hers own site and cannot see the other recruiting centers.
  * (project-redcap.org) (redcap.vanderbilt.edu)

REFERENCES:
- [Background] Northover JR, Wild JB, Braybrooke J, Blanco J. The epidemiology of cervical spondylotic myelopathy. Skeletal Radiol. 2012 Dec;41(12):1543-6. doi: 10.1007/s00256-012-1388-3. Epub 2012 Mar 17. PMID 22426774
- [Background] Kalsi-Ryan S, Karadimas SK, Fehlings MG. Cervical spondylotic myelopathy: the clinical phenomenon and the current pathobiology of an increasingly prevalent and devastating disorder. Neuroscientist. 2013 Aug;19(4):409-21. doi: 10.1177/1073858412467377. Epub 2012 Nov 30. PMID 23204243
- [Background] Nouri A, Tetreault L, Singh A, Karadimas SK, Fehlings MG. Degenerative Cervical Myelopathy: Epidemiology, Genetics, and Pathogenesis. Spine (Phila Pa 1976). 2015 Jun 15;40(12):E675-93. doi: 10.1097/BRS.0000000000000913. PMID 25839387
- [Background] Karadimas SK, Erwin WM, Ely CG, Dettori JR, Fehlings MG. Pathophysiology and natural history of cervical spondylotic myelopathy. Spine (Phila Pa 1976). 2013 Oct 15;38(22 Suppl 1):S21-36. doi: 10.1097/BRS.0b013e3182a7f2c3. PMID 23963004
- [Background] Kato S, Nouri A, Wu D, Nori S, Tetreault L, Fehlings MG. Comparison of Anterior and Posterior Surgery for Degenerative Cervical Myelopathy: An MRI-Based Propensity-Score-Matched Analysis Using Data from the Prospective Multicenter AOSpine CSM North America and International Studies. J Bone Joint Surg Am. 2017 Jun 21;99(12):1013-1021. doi: 10.2106/JBJS.16.00882. PMID 28632590
- [Background] Albert TJ, Vacarro A. Postlaminectomy kyphosis. Spine (Phila Pa 1976). 1998 Dec 15;23(24):2738-45. doi: 10.1097/00007632-199812150-00014. PMID 9879099
- [Background] Nori S, Shiraishi T, Aoyama R, Ninomiya K, Yamane J, Kitamura K, Ueda S. Muscle-Preserving Selective Laminectomy Maintained the Compensatory Mechanism of Cervical Lordosis After Surgery. Spine (Phila Pa 1976). 2018 Apr 15;43(8):542-549. doi: 10.1097/BRS.0000000000002359. PMID 28767627
- [Background] Parker SL, Godil SS, Shau DN, Mendenhall SK, McGirt MJ. Assessment of the minimum clinically important difference in pain, disability, and quality of life after anterior cervical discectomy and fusion: clinical article. J Neurosurg Spine. 2013 Feb;18(2):154-60. doi: 10.3171/2012.10.SPINE12312. Epub 2012 Nov 23. PMID 23176164
- [Background] Carreon LY, Glassman SD, Campbell MJ, Anderson PA. Neck Disability Index, short form-36 physical component summary, and pain scales for neck and arm pain: the minimum clinically important difference and substantial clinical benefit after cervical spine fusion. Spine J. 2010 Jun;10(6):469-74. doi: 10.1016/j.spinee.2010.02.007. Epub 2010 Apr 1. PMID 20359958
- [Background] Landriel Ibanez FA, Hem S, Ajler P, Vecchi E, Ciraolo C, Baccanelli M, Tramontano R, Knezevich F, Carrizo A. A new classification of complications in neurosurgery. World Neurosurg. 2011 May-Jun;75(5-6):709-15; discussion 604-11. doi: 10.1016/j.wneu.2010.11.010. PMID 21704941
- [Background] Kato S, Nouri A, Wu D, Nori S, Tetreault L, Fehlings MG. Impact of Cervical Spine Deformity on Preoperative Disease Severity and Postoperative Outcomes Following Fusion Surgery for Degenerative Cervical Myelopathy: Sub-analysis of AOSpine North America and International Studies. Spine (Phila Pa 1976). 2018 Feb 15;43(4):248-254. doi: 10.1097/BRS.0000000000002307. PMID 28658043
- [Background] Kawasaki M, Tani T, Ushida T, Ishida K. Anterolisthesis and retrolisthesis of the cervical spine in cervical spondylotic myelopathy in the elderly. J Orthop Sci. 2007 May;12(3):207-13. doi: 10.1007/s00776-007-1122-5. Epub 2007 May 31. PMID 17530371
- [Background] Shamji MF, Mohanty C, Massicotte EM, Fehlings MG. The Association of Cervical Spine Alignment with Neurologic Recovery in a Prospective Cohort of Patients with Surgical Myelopathy: Analysis of a Series of 124 Cases. World Neurosurg. 2016 Feb;86:112-9. doi: 10.1016/j.wneu.2015.09.044. Epub 2015 Sep 25. PMID 26409089
- [Background] White AA 3rd, Johnson RM, Panjabi MM, Southwick WO. Biomechanical analysis of clinical stability in the cervical spine. Clin Orthop Relat Res. 1975;(109):85-96. doi: 10.1097/00003086-197506000-00011. PMID 1132209
- [Background] Schizas C, Theumann N, Burn A, Tansey R, Wardlaw D, Smith FW, Kulik G. Qualitative grading of severity of lumbar spinal stenosis based on the morphology of the dural sac on magnetic resonance images. Spine (Phila Pa 1976). 2010 Oct 1;35(21):1919-24. doi: 10.1097/BRS.0b013e3181d359bd. PMID 20671589
- [Background] Wilson JRF, Badhiwala JH, Moghaddamjou A, Martin AR, Fehlings MG. Degenerative Cervical Myelopathy; A Review of the Latest Advances and Future Directions in Management. Neurospine. 2019 Sep;16(3):494-505. doi: 10.14245/ns.1938314.157. Epub 2019 Aug 26. PMID 31476852
- [Background] Woods BI, Hohl J, Lee J, Donaldson W 3rd, Kang J. Laminoplasty versus laminectomy and fusion for multilevel cervical spondylotic myelopathy. Clin Orthop Relat Res. 2011 Mar;469(3):688-95. doi: 10.1007/s11999-010-1653-5. PMID 21089002
- [Background] Badiee RK, Mayer R, Pennicooke B, Chou D, Mummaneni PV, Tan LA. Complications following posterior cervical decompression and fusion: a review of incidence, risk factors, and prevention strategies. J Spine Surg. 2020 Mar;6(1):323-333. doi: 10.21037/jss.2019.11.01. PMID 32309669
- [Background] Stromqvist B, Jonsson B, Fritzell P, Hagg O, Larsson BE, Lind B. The Swedish National Register for lumbar spine surgery: Swedish Society for Spinal Surgery. Acta Orthop Scand. 2001 Apr;72(2):99-106. doi: 10.1080/000164701317323327. No abstract available. PMID 11372956
- [Background] Stromqvist B, Fritzell P, Hagg O, Jonsson B; Swedish Society of Spinal Surgeons. The Swedish Spine Register: development, design and utility. Eur Spine J. 2009 Aug;18 Suppl 3(Suppl 3):294-304. doi: 10.1007/s00586-009-1043-4. Epub 2009 Jun 4. PMID 19495812
- [Background] Nurick S. The pathogenesis of the spinal cord disorder associated with cervical spondylosis. Brain. 1972;95(1):87-100. doi: 10.1093/brain/95.1.87. No abstract available. PMID 5023093
- [Background] Tetreault L, Nouri A, Kopjar B, Cote P, Fehlings MG. The Minimum Clinically Important Difference of the Modified Japanese Orthopaedic Association Scale in Patients with Degenerative Cervical Myelopathy. Spine (Phila Pa 1976). 2015 Nov;40(21):1653-9. doi: 10.1097/BRS.0000000000001127. PMID 26502097
- [Background] Rhee JM, Shi WJ, Cyriac M, Kim JY, Zhou F, Easley KA, Patel A. The P-mJOA: A Patient-derived, Self-reported Outcome Instrument for Evaluating Cervical Myelopathy: Comparison with the mJOA. Clin Spine Surg. 2018 Mar;31(2):E115-E120. doi: 10.1097/BSD.0000000000000591. PMID 29088009
- [Background] Young IA, Cleland JA, Michener LA, Brown C. Reliability, construct validity, and responsiveness of the neck disability index, patient-specific functional scale, and numeric pain rating scale in patients with cervical radiculopathy. Am J Phys Med Rehabil. 2010 Oct;89(10):831-9. doi: 10.1097/PHM.0b013e3181ec98e6. PMID 20657263
- [Background] Machino M, Imagama S, Ando K, Kobayashi K, Hida T, Ito K, Tsushima M, Matsumoto A, Tanaka S, Morozumi M, Ito K, Kato F, Nishida Y, Ishiguro N. Prospective Comparison of Age- and Sex-related Differences in Quantifiable 10-S Grip and Release and 10-S Step Test Results for Diagnosis of Cervical Spondylotic Myelopathy in 454 Patients With Cervical Spondylotic Myelopathy and 818 Asymptomatic Subjects. Spine (Phila Pa 1976). 2017 Apr 15;42(8):578-585. doi: 10.1097/BRS.0000000000001849. PMID 27513225
- [Background] Enoki H, Tani T, Ishida K. Foot Tapping Test as Part of Routine Neurologic Examination in Degenerative Compression Myelopathies: A Significant Correlation between 10-sec Foot-tapping Speed and 30-m Walking Speed. Spine Surg Relat Res. 2019 Jan 15;3(3):207-213. doi: 10.22603/ssrr.2018-0033. eCollection 2019. PMID 31440678
- [Background] Lofgren H, Osman A, Blomqvist A, Vavruch L. Sagittal Alignment After Laminectomy Without Fusion as Treatment for Cervical Spondylotic Myelopathy: Follow-up of Minimum 4 Years Postoperatively. Global Spine J. 2020 Jun;10(4):425-432. doi: 10.1177/2192568219858302. Epub 2019 Jun 26. PMID 32435562
- [Background] Tatter C, Fletcher-Sandersjoo A, Persson O, Burstrom G, Grane P, Edstrom E, Elmi-Terander A. Incidence and predictors of kyphotic deformity following resection of cervical intradural tumors in adults: a population-based cohort study. Acta Neurochir (Wien). 2020 Nov;162(11):2905-2913. doi: 10.1007/s00701-020-04416-4. Epub 2020 Jun 16. PMID 32556521
- [Background] Blackwelder WC. "Proving the null hypothesis" in clinical trials. Control Clin Trials. 1982 Dec;3(4):345-53. doi: 10.1016/0197-2456(82)90024-1. PMID 7160191
- [Background] White IR, Royston P, Wood AM. Multiple imputation using chained equations: Issues and guidance for practice. Stat Med. 2011 Feb 20;30(4):377-99. doi: 10.1002/sim.4067. Epub 2010 Nov 30. PMID 21225900
- [Derived] MacDowall A, Lofgren H, Edstrom E, Brisby H, Parai C, Elmi-Terander A. Comparison of posterior muscle-preserving selective laminectomy and laminectomy with fusion for treating cervical spondylotic myelopathy: study protocol for a randomized controlled trial. Trials. 2023 Feb 11;24(1):106. doi: 10.1186/s13063-023-07123-4. PMID 36765352